CLINICAL TRIAL: NCT03268668
Title: Thrombus Composition in Ischemic Stroke: Analysis of the Correlation With Plasma Biomarkers, Efficacy of Treatment, Etiology and Prognosis
Acronym: COMPO-CLOT
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JDS_2017_8
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Acute; Biological Specimen Banks; Biomarkers; Etiology; Prognosis
MeSH Terms: conditions — Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of thrombus that is responsible for stroke and blood sample — A blood sample (venous or arterial) of 10 ml will be made, on ethylene Diamine Tetra-Acetic (EDTA) tube (5 ml) and citrate (5 ml).Thrombus resulting from thrombectomy will be collected at the end of the procedure. The samples will be transferred to a biobank. Treatment efficacy, etiology and prognosis of patients will be assessed using the following criteria :
  A) TOAST score (etiology) B) TICI score (status of final recanalization) C) Extravasation of contrast agent on post-intervention CT (rupture of the blood-brain barrier :yes/no) D) Symptomatic haemorrhagic transformation corresponding to an increase > 4 of the NIHSS score due to a haemorrhagic transformation identified on brain imaging 24 hours after stroke E) Decreased NIHSS score by 8 points or NIHSS score = 0 24 hours after stroke (improved neurological status: yes/no) F) Modified RANKIN score (mRS) measured at 3 months evaluating neurological prognosis

SUMMARY:
The recent validation of thrombectomy in addition to thrombolysis with intravenous administration of alteplase suggests a major revolution in the management of acute strokes. This treatment option also opens up a new field of research, making possible the analysis of the clot responsible for intracranial occlusion. Indeed, in about 30% of the cases, the thrombectomy procedure makes it possible to retrieve either partially or completely the clot. Previous studies have analyzed the correlation between the composition of the thrombus and the etiology of stroke. Their discordant results do not yet make it possible to distinguish a particular profile of thrombus according to etiology. Other studies have shown a correlation between the proportion of red blood cells in a thrombus and the likelihood that it is visible in MRI or cerebral scanning. More recently, one study has demonstrated a correlation between the presence of lymphocytes in the thrombus and an atheromatous etiology.

The main limitations of these studies are the small number of patients included, the high variability of conservation protocols and the absence of plasma data, which does not allow for research on the correlation between clot composition and plasma biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Presenting with cerebral infarction following arterial occlusion
* Treated for mechanical thrombectomy (whether performed or not)
* Free, informed, and express consent of the patient or their relatives (emergency inclusion procedure)
* For retrospective patients: thrombus already collected (according to the center's usual practice or for another research project).

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ischemic stroke
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2027-07-12 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between the composition of the thrombus responsible for stroke, the plasma composition and the stroke characteristics (etiology, response to treatment, prognosis). | 3 months
  Since this is an observational, exploratory study that correlates laboratory data (eg for thrombus: fibrinolytic, pro-oxidant activity, eg for blood: plasma fibrinolysis markers, presence of factor Von Willebrand, etc.) and clinical data (characteristics of the stroke, including the TOAST etiological score, the TICI score (TICI = thrombolysis in cerebral infarction), the NIHSS score, etc.), there is no single primary endpoint.
  Clinical data will be collected up to 3 months after stroke (Rankin score).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Désilles, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (12):
- France (12):
  - CHU de Bordeaux, Bordeaux
  - CHU Caen, Caen
  - Chu Limoges, Limoges
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Lariboisière AP-HP, Paris
  - Centre hospitalier Sainte-Anne, Paris
  - Fondation Ophtalmologique A. de Rothschild, Paris
  - CHU de Rennes, Rennes
  - Hôpital Foch, Suresnes
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Meglio L, Desilles JP, Solonomenjanahary M, Labreuche J, Ollivier V, Dupont S, Deschildre C, Maacha MB, Consoli A, Lapergue B, Piotin M, Blanc R, Ho-Tin-Noe B, Mazighi M; compoCLOT study groupdagger. DNA Content in Ischemic Stroke Thrombi Can Help Identify Cardioembolic Strokes Among Strokes of Undetermined Cause. Stroke. 2020 Sep;51(9):2810-2816. doi: 10.1161/STROKEAHA.120.029134. Epub 2020 Aug 19. PMID 32811390